CLINICAL TRIAL: NCT06983678
Title: Neural Correlates and Behavioral Impact of Withdrawal-induced Hyperalgesia Among People Who Smoke With and Without Chronic Pain
Acronym: PRISM02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00117759; 1R01DA060859-01A1 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use; Chronic Pain
MeSH Terms: conditions — Tobacco Use; Chronic Pain | interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants with chronic pain - Smoking as usual fMRI session first followed by Abstinent fMRI (Experimental): Participants with chronic pain randomized to complete a smoking as usual fMRI session followed by an Abstinent fMRI session.
  Interventions: Behavioral: Smoking as usual fMRI session; Behavioral: Abstinent fMRI session
- Participants with chronic pain - Abstinent fMRI session first followed by Smoking as usual fMRI (Experimental): Participants with chronic pain randomized to complete an Abstinent fMRI session followed by a smoking as usual fMRI session.
  Interventions: Behavioral: Smoking as usual fMRI session; Behavioral: Abstinent fMRI session
- Participants without chronic pain - Smoking as usual fMRI session first followed by Abstinent fMRI (Experimental): Participants without chronic pain randomized to complete a smoking as usual fMRI session followed by an Abstinent fMRI session.
  Interventions: Behavioral: Smoking as usual fMRI session; Behavioral: Abstinent fMRI session
- Participants without chronic pain - Abstinent fMRI session first followed by Smoking as usual fMRI (Experimental): Participants without chronic pain randomized to complete an Abstinent fMRI session followed by a smoking as usual fMRI session.
  Interventions: Behavioral: Smoking as usual fMRI session; Behavioral: Abstinent fMRI session

INTERVENTIONS:
Behavioral: Smoking as usual fMRI session — Participants in this condition will continue smoking as usual prior to the fMRI session
Behavioral: Abstinent fMRI session — Participants in this condition will be asked to abstain from smoking or using any other tobacco products for 24 hours prior to the fMRI session

SUMMARY:
Individuals with chronic pain are more likely to smoke cigarettes and have more difficulty quitting smoking than the general population, in part because withdrawal from smoking can lead to temporary increases in pain. This research will examine how smoking withdrawal changes the way the brain processes pain, and whether these withdrawal-related changes interfere with the ability to stop smoking. The results of this research will provide important information that can be used to guide the development of interventions to help people with chronic pain who smoke cigarettes to quit smoking and improve their health.

DETAILED DESCRIPTION:
Eligible participants will complete an initial in-person screening session in which eligibility is confirmed and baseline pain and smoking measures are collected, followed by a sensory testing and training session, in which participants are introduced to the mock MRI scanner and familiarized with the thermal pain stimulation and psychophysiological rating procedures. Participants will then complete two fMRI sessions using a within-subjects, crossover design, with one scan following 24-hrs abstinence from smoking, and the other following smoking as usual. Both fMRI sessions will be identical other than the smoking instructions prior to the scan. During each scan, participants will complete experience and provide ratings to painful heat stimuli. Before and after scanning, participants will complete measures of craving, withdrawal, and current pain level. After completion of the scanning sessions, participants will return to the lab for a baseline visit prior to beginning the abstinence test. During that session, they will have software installed on their smartphone for ecological momentary assessment (EMA), and they will be trained in the procedures for biochemical verification of abstinence. They will then complete 3 days of baseline EMA, during which participants are prompted at 5 random times throughout the day, and once in the evening, to answer questions about their pain, smoking urge, and recent smoking. They will then continue EMA while attempting to abstain from smoking during the 1-week abstinence test. During the abstinence test, each day of abstinence is reinforced with money using a descending schedule. Participants will provide breath samples over video during this week using equipment provided by the lab in order to verify abstinence from smoking. At the conclusion of the study, participants will return to the lab for a final visit to return all equipment.

ELIGIBILITY:
Inclusion Criteria:

1. History of chronic non-cancer low back pain with duration ≥ 6 months OR no history of chronic pain;
2. age 21-65;
3. smoking of at least 10 cig/day for > 2 years;
4. have an iPhone or Android smartphone capable of running the EMA software

Exclusion Criteria:

1. pain complaint specifically due to cancer, rheumatoid arthritis, or complex regional pain syndrome;
2. actively taking steps to quit smoking;
3. inability to attend all required experimental sessions;
4. significant health problems, such as chronic hypertension, emphysema, seizure disorder, history of significant heart problems;
5. conditions that would make MRI scanning unsafe (e.g., metal implants, claustrophobia)
6. use of opioids within the past 90 days
7. past year alcohol or substance use disorder
8. positive urine test for illegal drugs (other than marijuana);
9. daily use of alcohol or marijuana;
10. lifetime history of psychotic disorder, or current unstable psychiatric disorder;
11. regular use of non-cigarette tobacco products or electronic cigarettes;
12. major surgery within the past 6 months or planned surgery within the timeframe of the study;
13. breath alcohol level > 0.0 (participants failing for BAL will be allowed to rescreen once);
14. recently quit smoking for > 3 days;
15. pregnancy or planning to become pregnant;
16. any factors that at the discretion of the investigators would adversely affect the participant or integrity of the study (e.g., ongoing legal action or disability claim regarding pain, uncontrolled psychiatric disorder, head/neck injury, use of certain medications)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity ratings to high heat vs neutral temperatures | Measured at each fMRI session (up to 1.5 hours)
  Participants will rate their current pain intensity following each of the heat stimulus blocks during the fMRI scans. Pain intensity is measured on a 0-10 visual analogue scale, with higher scores indicating greater pain.
Activation of the inferior frontal gyrus (IFG) | Measured at each fMRI session (up to 1.5 hours)
  % signal change in response to the contrast of high heat vs rest will be extracted from right and left IFG
Resting state functional connectivity with the IFG | Measured at each fMRI session (up to 1.5 hours)
  Fisher-Z transformed correlation maps of connectivity with the IFG will be evaluated within a subcortical mask including the caudate and thalamus
Time to lapse | Measured daily during the 1-week abstinence test
  The number of days of continuous, biochemically verified abstinence prior to smoking
Daily pain ratings | Measured with daily EMA prompts for 10 days
  Mean pain ratings during the initial days of abstinence will be examined as a function of chronic pain status, assessed at baseline
Daily withdrawal symptoms | Measured with daily EMA prompts for 10 days
  Daily withdrawal symptoms will be assessed over EMA using the Minnesota Smoking Withdrawal Scale. Mean withdrawal symptoms during the initial days of abstinence will be examined as a function of chronic pain status, assessed at baseline
Fluctuations in pain ratings vs smoking urge | Measured 5 times per day with random EMA prompts for 10 days
  Fluctuations in pain ratings will be examined to determine their association with level of smoking urge
Fluctuations in pain ratings vs number of cigarettes smoked | Measured 5 times per day with random EMA prompts for 10 days
  Fluctuations in pain ratings will be examined to determine their association with number of cigarettes smoked between each assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Sweitzer, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke North Pavilion, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No